CLINICAL TRIAL: NCT04356495
Title: Randomized Trial to Evaluate the Safety and Efficacy of Outpatient Treatments to Reduce the Risk of Worsening in Individuals With COVID-19 With Risk Factors (COVERAGE France)
Brief Title: Trial of COVID-19 Outpatient Treatment in Individuals With Risk Factors for Aggravation
Acronym: COVERAGEFrance
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: University of Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2020/12
Record Dates: First submitted 2020-04-11; First posted 2020-04-22 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Corona Virus Infection; Sars-CoV2
Keywords: Corona virus; Sars-CoV2; telmisartan; ciclesonide; interferon β-1b
MeSH Terms: conditions — Coronavirus Infections | interventions — Vitamins; Telmisartan; ciclesonide

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, controlled clinical trial with for each drug :
  * A safety study pilot phase.
  * An efficacy study phase. The data collected during the pilot phase, combined with new external data that emerged during the period, will be used to position treatments for the efficacy phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vitamins (Sham Comparator): Patients in this arm will receive a vitamin supplement ("AZINC forme et vitalité®") during 10 days
  Interventions: Dietary Supplement: Vitamins
- Telmisartan (Experimental): Patients in this arm will receive Telmisartan (Micardis® 20 mg) during 10 days
  Interventions: Drug: Telmisartan
- Ciclesonide (Experimental): Patients in this arm will receive ciclesonide (Alvesco® 160 µg ) during 10 days
  Interventions: Drug: Ciclesonide
- interferon β-1b (Experimental): Patients in this arm will receive interferon β-1b (Extavia® 9,6 MUI/300 µg ) during 5 days
  Interventions: Drug: interferon β-1b

INTERVENTIONS:
Dietary Supplement: Vitamins — 2 tablets daily from the first day (day 0) to day 9
  Arms: Vitamins
Drug: Telmisartan — 1 tablet daily from the first day (day 0) to day 9
  Arms: Telmisartan
Drug: Ciclesonide — 2 puffs twice a day in an inhalation chamber from the first day (day 0) to day 9
  Arms: Ciclesonide
Drug: interferon β-1b — A 10-minute nebulization, once a day, from the first day (day 0) to day 4, of 9.6 MIU / 300 µg of IFN-β-1b (EXTAVIA®) diluted in 2 mL of water
  Arms: interferon β-1b

SUMMARY:
In adults with COVID-19 without criteria for hospitalization or oxygen therapy but with risk factors for aggravation, early treatment may avoid hospitalization, indication for oxygen therapy or death. No treatment is currently validated for this indication.

DETAILED DESCRIPTION:
COVERAGE France is Multicenter, randomized, controlled clinical trial with for each drug :

* A safety study pilot phase.
* An efficacy study phase. The data collected during the pilot phase, combined with new external data that emerged during the period, will be used to position treatments for the efficacy phase.
* Pilot phase will evaluate the tolerance of experimental treatments for drugs given for the first time ("first in home-based care") in ambulatory individuals with COVID-19 with aggravating risk factors.
* Efficacy Phase: To estimate the effectiveness of experimental ambulatory treatments, compared to vitamin supplementation, in reducing the risk of hospitalization, oxygen therapy indication or death in ambulatory individuals with COVID-19 with aggravating risk factors.

The trial is a national platform with the vocation to open as many centers as possible, subject to criteria set by the Scientific Advisory Board.

ELIGIBILITY:
Inclusion Criteria:

* Clinical picture suggestive of COVID-19 dated 7 days or less.
* Positivity of a test proving an acute SARS-CoV-2 infection, according to current recommendations.
* Absence of criteria for hospitalization or oxygen therapy according to current recommendations.
* Age :

  * greater than or equal to 60 years of age without any risk factor
  * or between 50 and 59 years of age and the presence of at least one of the following risk factors :

    * Arterial hypertension under treatment (all stages)
    * Obesity (BMI ≥30 kg/m2)
    * Diabetes under treatment (all types)
    * Ischemic heart disease (all stages)
    * Heart failure (all stages)
    * Stroke History
    * Chronic Obstructive Pulmonary Disease (all stages)
    * Stage 3 chronic renal failure (30 ≤ Estimated GFR < 60 mL/min/1.73 m²)
    * Malignancies (solid tumours or blood malignancies) that are progressive or were diagnosed less than 5 years ago.
    * Immunodeficiency
* of therapeutic origin (solid organ transplant or hematopoietic stem cell transplant, cancer chemotherapy, immunosuppressive therapy, corticosteroids > 15 mg/d of prednisone equivalent taken for at least 2 months);
* HIV infection with CD4<200/mm3.
* Valid, ambulatory person, fully able to understand the issues of the trial
* Beneficiary of a Social Security scheme
* Signed informed consent

Exclusion Criteria:

* Asymptomatic person
* Inability to make a decision to participate (dementia, person under legal protection, curatorship or guardianship)
* Ongoing illness or chronic treatment contraindicated by taking one of the trial drugs.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
Pilot Phase: Proportion of participants who had a Grade 3 or 4 adverse event | From inclusion (day0) to day 14
Efficacy phase: Death | From inclusion (day0) to day 14
  Proportion of participants with an occurrence of death
Efficacy phase: oxygen therapy | From inclusion (day0) to day 14
  Proportion of participants who had an indication for oxygen therapy
Efficacy phase: hospitalization | From inclusion (day0) to day 14
  Proportion of participants who had an indication for hospitalization

SECONDARY OUTCOMES:
Proportion of hospitalizations, overall and by cause, in each group | From inclusion (day0) to day 28
Death and causes of death | From inclusion (day0) to day 28
  Proportion of deaths, overall and by cause, in each group
Proportion of intensive care hospitalizations, overall and by cause, in each group | From inclusion (day0) to day 28
Proportion of participants with negative SARS-CoV-2 RT-PCR | day 7
Haematological markers evolution | from inclusion (day 0) to day 7
  Evolution of Haematological markers in each group : Complete Blood Count, prothrombin level, INR
Inflammatory markers evolution | from inclusion (day 0) to day 7
  Evolution of Inflammatory markers in each group : PCT, CRP
Adverse events | from inclusion (day 0) to day 28
  Number and proportion of grade 1,2,3,4 adverse events in each group
Adverse reactions | from inclusion (day 0) to day 28
  Number and proportion of grade 1,2,3,4 adverse events in each group
Acceptability of the treatment | from inclusion (day 0) to day 10
  Acceptability of the treatment by participant will be assessed with an interview
Antibiotic consumption | from inclusion (day 0) to day 28
  Proportion of participants who received at least one day of antibiotic therapy
Oxygen saturation worsening | from inclusion (day 0) to day 28
  Proportion of participants who experienced a worsening of oxygen saturation
protocol follow-up | from inclusion (day 0) to day 10
  Proportion of participants who completed the prescribed protocol treatment

CONTACTS AND LOCATIONS:
Overall Officials: Denis MALVY, Pr, Principal Investigator — University Hospital, Bordeaux; Xavier ANGLARET, Dr, Study Director — Inserm 1219; Laura RICHERT, Dr, Study Chair — University Hospital, Bordeaux
Locations (7):
- France (7):
  - Bordeaux university Hospital, Bordeaux
  - CHU de Dijon-Bourgogne, Dijon
  - CHU de Montpellier, Montpellier
  - CHRU de Nancy, Nancy
  - Groupe hospitalier Paris Saint Joseph, Paris
  - CNGE, Paris
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Garcia G, Labrouche-Colomer S, Duvignaud A, Clequin E, Dussiau C, Tregouet DA, Malvy D, Prevel R, Zouine A, Pellegrin I, Goret J, Mamani-Matsuda M, Dewitte A, James C. Impaired balance between neutrophil extracellular trap formation and degradation by DNases in COVID-19 disease. J Transl Med. 2024 Mar 7;22(1):246. doi: 10.1186/s12967-024-05044-7. PMID 38454482
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] Duvignaud A, Lhomme E, Pistone T, Onaisi R, Sitta R, Journot V, Nguyen D, Peiffer-Smadja N, Cremer A, Bouchet S, Darnaud T, Poitrenaud D, Piroth L, Binquet C, Michel JF, Lefevre B, Lebeaux D, Lebel J, Dupouy J, Roussillon C, Gimbert A, Wittkop L, Thiebaut R, Orne-Gliemann J, Joseph JP, Richert L, Anglaret X, Malvy D; COVERAGE study group. Home Treatment of Older People with Symptomatic SARS-CoV-2 Infection (COVID-19): A structured Summary of a Study Protocol for a Multi-Arm Multi-Stage (MAMS) Randomized Trial to Evaluate the Efficacy and Tolerability of Several Experimental Treatments to Reduce the Risk of Hospitalisation or Death in outpatients aged 65 years or older (COVERAGE trial). Trials. 2020 Oct 13;21(1):846. doi: 10.1186/s13063-020-04619-1. PMID 33050924